CLINICAL TRIAL: NCT06588725
Title: Brief Interventions to Improve Behavior Outcomes and Prevent Cavities
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Seth Scholer, Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 241240
Record Dates: First submitted 2024-08-07; First posted 2024-09-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-10

CONDITIONS: Parenting; Cavity, Dental; Child Behavior
MeSH Terms: conditions — Dental Caries; Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child behavior management - free resources (Experimental): Two minutes of education about child behavior management coupled with free resources.
  Interventions: Behavioral: Play Nicely
- Child behavior management - handbook (Experimental): Two minutes of education about child behavior management coupled with free resources and a handbook
  Interventions: Behavioral: Play Nicely
- Cavity Prevention (Experimental): Two minutes of education about how to prevent cavities coupled with a 2 page handout.
  Interventions: Behavioral: Cavity Prevention Handout

INTERVENTIONS:
Behavioral: Play Nicely — Multimedia tool and handbook designed to educate parents about healthy discipline strategies.
  Arms: Child behavior management - free resources; Child behavior management - handbook
Behavioral: Cavity Prevention Handout — Two page handout with information about how to prevent cavities.
  Arms: Cavity Prevention

SUMMARY:
The investigators will study brief educational interventions designed to address childhood behavior problems and prevent cavities.

DETAILED DESCRIPTION:
The investigators will study brief educational interventions designed to address childhood behavior problems and prevent cavities. Participants will be parents of children, ages 9 months to 3 years, presenting with their child for a well child visit. Parent/child dyads will be randomized into three different groups: Group 1 will be introduced to an online educational intervention to address childhood behavior problem, Group 2 will be introduced to a printed educational intervention to address childhood behavior problems, and Group 3 will be introduced to an educational intervention to prevent cavities. Study procedures will include 1) the educational intervention in the examination room before the clinic visit, 2) a brief survey immediately after the clinic visit and 3) a brief survey in 2-4 months sent via REDCap, and 4) follow up health and insurance records related to the study interventions.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 9 month to 3 year old children.

Exclusion Criteria:

-

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Child behavior problems | 3 years, or until the end of the study.
  We will review the medical chart for the following outcomes: Number of participants with child behavior problems; referral to mental/behavioral health provider; use of psychotropic medications.
Cavity-related outcomes | 3 years, or until the end of the study.
  We will review the medical chart and dental records for cavity related outcomes including number of children with cavities, fillings, and crowns.

SECONDARY OUTCOMES:
Planned change to care for behavioral health | Same day as enrollment, for 3 years or until the end of the study.
  The survey will ask parents about planned change to care for child's behavioral health and ask about whether the parent feels that they have the resources to address behavioral needs.
Planned change to prevent cavities | Same day as enrollment, for 3 years or until the end of the study.
  The survey will ask parents about planned change to prevent cavities and ask about whether the parent feels that they have the resources to prevent cavities.
Report on helpfulness of interventions | 2-4 months after enrollment, for 3 years or until the end of the study.
  The survey will ask parents whether the information they received at the well visit was helpful and what, if anything, they are doing differently to address behavioral health or to prevent cavities.

CONTACTS AND LOCATIONS:
Overall Officials: Seth J Scholer, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Children's Primary Care One Hundred Oaks, Nashville, Tennessee, United States